CLINICAL TRIAL: NCT06538844
Title: Albumin for Patients With Acute Large Vessel Occlusive Stroke Undergoing Endovascular Reperfusion Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARISE
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-08

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Human albumin treatment group (Experimental)
  Interventions: Drug: Intravenous infusion of human albumin
- Placebo group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Intravenous infusion of human albumin — Administer 0.5g/kg of 25% human albumin intravenously as soon as possible within 60 minutes after randomization. And administer 0.5g/kg of 25% ALB intravenously every day on the second, third, and fourth days after randomization.
  Arms: Human albumin treatment group
Drug: Saline — Equivalent volume of isotonic saline control
  Arms: Placebo group

SUMMARY:
The objective of this study is to evaluate the effectiveness and safety of endovascular therapy combined with 25% human albumin in the treatment of acute large vessel occlusive stroke.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide, 85% of which are acute ischemic strokes (AIS). Neuronal death is the primary pathological manifestation of acute ischemic stroke (AIS). Preclinical studies have revealed that neuroprotective agents can reduce neuronal damage and improve neurological outcomes in experimental animals. However, over the past 40 years, clinical translation of neuroprotective drugs has consistently failed. In 2015, with the publication of five randomized controlled trials (RCTs) on thrombectomy for anterior circulation, there was sufficient evidence-based support for thrombectomy in large vessel occlusion of the anterior circulation, ushering us into a new era of AIS treatment - the era of efficient reperfusion therapy. In this context, neuroprotective therapy should be re-examined as an adjunctive approach to reperfusion therapy.

Albumin, the predominant plasma protein synthesized primarily in the liver, possesses various biochemical properties that are expected to confer a neuroprotective effect following acute ischemic stroke.

This study is a multi-center, randomized, double-blind, placebo-controlled clinical study, focusing on patients with acute large vessel occlusive stroke. It aims to investigate the effectiveness and safety of albumin as an adjunctive treatment to endovascular therapy compared with placebo in reducing infarct volume, improving long-term functional outcomes, and daily living activities of patients with acute ischemic stroke in the era of reperfusion therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years;
2. Anterior circulation acute ischemic stroke, with acute occlusion of the responsible vessel located in the intracranial segment of the internal carotid artery, or the M1 or M2 segment of the middle cerebral artery;
3. National Institute of Health Stroke Scale (NIHSS) score ≥6;
4. Modified Rankin Scale (mRS) score ≤1 before onset of the disease;
5. Alberta Stroke Program Early CT Score (ASPECTS) ≥3 points;
6. Ischemic-core volume ≤100ml;
7. Patient treatable within 24 hours of symptom onset. Symptoms onset is defined as point in time the patient was last seen well (at baseline) if patients are unable to provide a reliable history or the point in time when symptoms have started if patients can provide a reliable history. Treatment start is defined as groin puncture.;
8. Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

1. Evidence of intracranial hemorrhage (intracerebral hematoma (ICH), subarachnoid hemorrhage (SAH), epidural hemorrhage, acute or chronic subdural hematoma (SDH)) on the baseline CT or MRI scan；
2. History of congenital or acquired bleeding disorders, coagulation factor deficiency diseases, thrombocytopenic diseases, etc;
3. Anticipated difficulty in completing endovascular treatment due to vascular tortuosity;
4. Known severe allergy (more severe than skin rash) to contrast agents uncontrolled by medications;
5. Pregnancy, breastfeeding；
6. An episode or exacerbation of congestive heart failure from any cause in the past 6 months;
7. History of heart valve disease complicated by congestive heart failure within the past 6 months；
8. Cardiac surgery with thoracotomy (eg coronary artery bypass grafting or valve replacement surgery) within the past 6 months；
9. Acute myocardial infarction in the past 6 months;
10. Signs or symptoms of acute myocardial infarction upon admission, including electrocardiographic findings；
11. Elevated serum troponin concentration upon admission (>0.1 μg/L) ；
12. Acute arrhythmia (including any tachycardia or bradycardia) with hemodynamic instability (systolic blood pressure <100 mm Hg) upon admission；
13. Acute or chronic lung diseases requiring long-term or intermittent oxygen therapy；
14. Findings on physical examination of any of the following abnormalities: (1) Jugular venous distension (jugular venous pulsation >4 cm above the sternal angle); (2) Resting tachycardia due to congestive heart failure (heart rate > 100 per/min); (3) Third heart sound; (4) Abnormal hepatic jugular venous reflux; (5) Pitting edema of the lower extremities attributable to congestive heart failure or without apparent cause; (6) Rales in both lungs; (7) Or evidence of pulmonary edema, pleural effusion, or pulmonary vascular redistribution on chest X-ray；
15. Known recent or current serum creatinine exceeding 1.5 times the upper limit of normal, or estimated glomerular filtration rate (eGFR) < 60 mL/min;
16. Refractory hypertension that is difficult to control by medication (defined as systolic blood pressure > 220 mmHg, or diastolic blood pressure > 110 mmHg);
17. Severe chronic anemia (hemoglobin < 75 g/L);
18. History of albumin allergy or known allergy to albumin;
19. Patients with severe mental disorders or dementia who are unable to cooperate in completing informed consent and follow-up content;
20. The expected survival time is less than 90 days (such as comorbidity with malignant tumor or severe systemic diseases etc.);
21. Patients who have participated in other interventional clinical studies within 30 days prior to randomization or are currently participating in other interventional clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Changes in infarction volume from Day 5 to baseline. | From 5 days after surgery to baseline

SECONDARY OUTCOMES:
Early neurological improvement within 24 hours | within 24 hours
  Decrease in National Institute of Health stroke scale (NIHSS) score of ≥8 or NIHSS score of 0-2 within 24 hours. NIHSS scores range from 0 to 42, with higher scores indicating greater neurologic deficit
NIHSS score at 24 hours | at 24 hours
  National Institutes of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating greater neurologic deficit
Proportion of successful reperfusion (mTICI 2b/3) | immediate postoperative
  mTICI denotes modified Treatment in Cerebral Ischemia classification, with scores ranging from 0 (no flow) to 3 (normal flow)
NIHSS score at 5 days | at 5 days
  National Institutes of Health Stroke Scale (NIHSS)
Proportion of patients with functional independence (mRS 0-1) at 90 days | at 90 days
  Scores on the modified Rankin scale range from 0 to 6, with higher scores indicating greater disability
Proportion of patients with functional independence (mRS 0-2) at 90 days | at 90 days
  Scores on the modified Rankin scale range from 0 to 6, with higher scores indicating greater disability
Proportion of patients with Barthel Index of 95-100 at 90 days | at 90 days
European quality of Life-5 Dimensions (EQ-5D) at 90 days | at 90 days
  EQ-5D is a standardized instrument for the measurement of health status. Scores range from -0.33 to 1.00, with higher scores indicating a better quality of life
Incidence of Symptomatic intracerebral hemorrhage (ICH) Within 24 Hours | within 24 hours
Incidence of Intracerebral hemorrhage within 24 Hours | within 24 hours
Neurological deterioration within 24 hours | within 24 hours
  NIHSS score increased by ≥4 points within 24 hours.
Incidence of New-onset atrial fibrillation within 5 days | within 5 days
Incidence of Pulmonary edema or congestive heart failure within 5 days | within 5 days
Incidence of Intracerebral hemorrhage within 5 days | within 5 days
Incidence of Symptomatic intracerebral hemorrhage (ICH) Within 5 days | within 5 days
Incidence of Decompressive craniectomy within 7 days | within 7 days
Death within 90 days | within 90 days
Number of participants who experience adverse events (AEs) | within 90 days
Number of participants who experience serious adverse events (SAEs) | within 90 days

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Maanshan People's Hospital, Ma’anshan, Anhui
  - Suzhou Municipal Hospital of Anhui Province, Suzhou, Anhui
  - Luoyang Central Hospital Affiliated to Zhengzhou University, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - First People's Hospital of Zhengzhou City, Zhengzhou, Henan
  - Xihua County People's Hospital, Zhoukou, Henan
  - Northern Jiangsu People's Hospita!, Yangzhou, Jiangsu
  - Liaocheng Third People's Hospital, Liaocheng, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Dong X, Chu X, Ma Z, Yi T, Wen C, Liu Y, Sun J, Xu J, Li W, Yang L, Wang B, Shi L, Li J, Zhang X, Li C, Chen W, Li C, Wu D, Hou C, Zhou C, Li M, Xu Y, Wu C, Ji X. Albumin for patients with acute large-vessel occlusive stroke undergoing endovascular therapy (ARISE): the protocol of a randomized double-blind trial. Front Neurol. 2025 Jul 18;16:1570184. doi: 10.3389/fneur.2025.1570184. eCollection 2025. PMID 40757028